CLINICAL TRIAL: NCT02171884
Title: Study of the Impact of Freezing-thawing Procedures and the Prolonged Culture of Embryos on Epigenetic Regulation in Humans
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: FAUQUE DB 2013
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Assisted Reproductive Technology; Freezing/Thawing Procedure; Prolonged Culture Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Group E1: Singletons born following ART via IVF/ICSI (short culture)
  Interventions: Other: Sample of cord blood; Other: Sample of placenta
- Group EC1: Singletons born following ART via IVF/ICSI and freezing-thawing of the embryo
  Interventions: Other: Sample of cord blood; Other: Sample of placenta
- Group T1: Singletons conceived naturally
  Interventions: Other: Sample of cord blood; Other: Sample of placenta
- Group E2: Singletons born following ART with IVF/ICSI (prolonged culture)
  Interventions: Other: Sample of cord blood; Other: Sample of placenta

INTERVENTIONS:
Other: Sample of cord blood
Other: Sample of placenta

SUMMARY:
For this project, 4 groups of 38 infants have been created so as to evaluate the impact of Assisted-Reproduction Technology (ART) and more particularly the two procedures classically used in ART: the freezing/thawing of embryos and prolonged embryo culture (five days of culture in appropriate in vitro conditions to allow development of the embryo) in contrast with shorter culture of only two days.

Participation consists in accepting samples to be taken at the birth of the infant:

1. from the umbilical cord.
2. from the placenta.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent,
* Patients with national health insurance cover,
* Maternal age at conception between 20 and 43 years,
* Paternal age at conception between 18 and 50 years,
* Singleton pregnancy

Exclusion Criteria:

---Maternal disease:

* pulmonary, cardiac
* renal and metabolic diseases (including type 1 and 2 diabetes prior to the pregnancy)
* systemic inflammatory diseases
* hypertension
* neurological diseases
* chronic hepatitis B or C
* HIV infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 4 groups of infants:
  * conceived naturally
  * born following ART with IVF/ICSI (short culture)
  * born following ART with IVF/ICSI and freezing/thawing of the embryo
  * born following ART with IVF/ICSI (prolonged culture)
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Analysis of the expression of several genes subjected to imprinting (H19, IGF2, IGF2R, MEST, PEG3, SNRPN, IGF2, KCNQ1, GRB10 and PLAGL1) | Baselines
  DNA / RNA extraction
Analysis of the expression of 3 transposable elements (HERV-K, LINE-1 and ALU) | Baselines
  DNA / RNA extraction
Level of methylation and the level of expression of Genomic Imprinting (GI) and Transposable Elements (TE) | Baselines
  DNA / RNA extraction

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de BESANCON, Besançon
  - CHU de DIJON, Dijon